CLINICAL TRIAL: NCT04575974
Title: Combined Lifestyle Factors in Adolescence and Later Persistent Musculoskeletal Pain in Young Adulthood: Prospective Analyses From the HUNT Study
Brief Title: Lifestyle in Adolescence and Persistent Musculoskeletal Pain in Young Adulthood
Status: Completed | Type: Observational
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Britt Elin Øiestad, Accociate Professor, Oslo Metropolitan University
Other Study IDs: 2019/517B
Record Dates: First submitted 2020-09-08; First posted 2020-10-05 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Musculoskeletal Pain
Keywords: Musculoskeletal pain; Adolescence, young adulthood; Lifestyle; Risk factor
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents 13-19 years: All adolescents between 13-19 years of age in North Trøndelag county were invited to participate in HUNT 3 and followed up after 11 years.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Experiencing an episode of musculoskeletal (MSK) pain in young age significantly increases the risk of developing MSK pain later in life. Consequently, knowledge on modifiable risk factors early in life is needed. In this prospective cohort study, data from the population-based Nord-Trøndelag Health Study (HUNT) will be used to investigate whether a combination of lifestyle factors in adolescence is associated with persistent MSK pain in young adulthood.

DETAILED DESCRIPTION:
There is need for knowledge on modifiable risk factors for MSK pain in young ages to better target treatment and preventive. A combination of lifestyle factors has been associated with several health issues including MSK pain in adults, but has to the best of our knowledge not previously been investigated as a risk factor for MSK pain in the youth.

OBJECTIVE The objective of this study is to investigate whether a combination of lifestyle factors in adolescence is associated with later persistent MSK pain in young adulthood. Lifestyle factors will be assessed by combing levels of physical activity, sleep problems, fruit/vegetable consumption, alcohol consumption, use of drugs and smoking.

The analysis will be conducted in a sample of adolescents with MSK pain, and in a sample of adolescents without MSK pain in the first survey, separately.

STUDY DESIGN AND PLAN This study will be a prospective cohort study using data from the large population-based Nord Trøndelag Health Study (HUNT). Data from YoungHUNT3 (2006-2008) and HUNT4 (2017-2019) will be used, including the same participants examined With 11-year follow-up. The data in Young-HUNT 3 was collected through questionnaires, interviews and measurements during school time. Adolescents, who did not attend school, received an invitation to participate by mail. The outcome data was obtained by electronic questionnaire or paper from HUNT 4.

EXPOSURE VARIABLE A combined lifestyle variable will be composed based on scorings in the lifestyle variables physical activity level, sleep problems, fruit/vegetable consumption, alcohol consumption, drug use and smoking level from Young-HUNT3, which will all be categorized as healthy/ unhealthy (as defined below). The combined lifestyle variable will be arranged with 0/1 unhealthy lifestyle factors present as the reference category, and 2 factor, 3 factors and ≥4 unhealthy lifestyle factors present as the other categories. The combined variable will be investigated with different thresholds of alcohol consumption.

* Physical activity level: less than 2-3 days a week with sports or exercise is classified as a unhealthy level.
* Sleep problems is measured by two questions; one of whether the adolescents have problems falling asleep at night and one of whether the adolescents wake up early and have problems falling asleep again. Answering "often" or "almost every night" on one or both of these questions is classified as unhealthy.
* Fruit / vegetables consumption is measured by questions of consumption frequency. Answering "several times a day" on both questions will be considered a sufficient consumption.
* Alcohol consumption is measured by a question of whether the participants have ever tried to drink alcohol, and a question of whether the participants have ever been drinking so much that they have felt intoxicated (drunk). Those who have never tried drinking alcohol or have been intoxicated ≤10 times will be classified as healthy. Reporting >10 intoxications will be classified as unhealthy.
* Use of drugs: those who answer that they have tried hash, marijuana or other drugs will form the unhealthy group.
* Smoking will be dichotomized with no smokers in the healthy group and daily and occasional smokers in the unhealthy group. Previously smokers will be included in the no smoking group.

CONFOUNDING FACTORS

Background factors

* Sex
* Age
* Perceived family economic

Health factors

* Psychological distress, measured by the Symptom Checklist-5.
* Other chronic diseases, including asthma, diabetes, migraine and/or epilepsy
* Pain impact on daily activities at baseline (in the analyses of the sample with MSK pain at baseline only)
* Number of pain sites at baseline (in the analyses of the sample with MSK pain at baseline only)

(Additional analyses will be conducted with adjustment for BMI, measured by kg/m2).

ANALYSIS METHODS Statistical tests will be two-sided, and p-values <0.05 will be considered statistically significant. P-value and the 95% confidence intervals will be reported. All continuous variables will be investigated for normality through histograms and QQ-plots. Normally distributed descriptive data of study participant will be presented with means and standard deviations (SD), skewed data will be presented with median and ranges and categorical data will be presented as counts and percentages. The analysis will be conducted with STATA statistical software system.

Missing data:

For missing data on the exposure variable and confounding factors, multiple imputation will be considered. Variables with more than 20% missing data will be excluded. Participants with missing outcome data will be excluded from the analyses. Characteristics of the individuals lost to follow-up will be compared to characteristics of responders at follow-up.

Incidence and prevalence:

The prevalence and incidence rate of MSK pain will be presented.

Logistic regression:

Logistic regression will be used to investigate the association between combined lifestyle factors in adolescence and persistent MSK pain in young adulthood. The combined lifestyle factor variable will be investigated with different thresholds of alcohol consumption. The associations will be investigated in unadjusted and adjusted analyses. The adjusted analyses will be conducted first with adjustment for background factors, second with adjustment for background factors and health factors. There will be conducted additional analyses with adjustment for BMI (kg/m2). The results will be reported as odds ratios (ORs) with 95% confidence intervals.

Sub-group analyses:

There will be conducted subgroup analyses for girls and boys separately, if there is a sufficient number of participants.

ELIGIBILITY:
Inclusion Criteria:

* Respondents in Young-HUNT 3

Exclusion Criteria:

* Participants reporting juvenile arthritis
* Participants ≥ 20 years in Young-HUNT3

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents (13-19 years) from Nord-Trøndelag in Norway.
Sampling Method: Non-Probability Sample
Enrollment: 8562 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Persistent musculoskeletal pain lasting 3 months or more during the last year | 1 year (measured 11 years after baseline)
  The outcome was measured by the question: "In the last year, have you had pain or stiffness in muscles or joints that has lasted at least 3 consecutive months?" The responses were dichotomised into yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Britt Elin Øiestad, PhD, Principal Investigator — Oslo Metroplitan University

IPD SHARING:
Plan to Share IPD: No
Data are available from the HUNT database, but restrictions apply to the availability of these data, which were used under license for the current study.